CLINICAL TRIAL: NCT00987246
Title: Study on the Efficacy of LAS41005 Compared to Placebo and to LAS106521 in the Treatment of Actinic Keratosis Grade I to II
Brief Title: Study on the Efficacy of LAS41005 in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H 1005 6002 - 0702; EudraCT: 2007-003889-18
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; AK; NMSC; Combination
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAS41005 (Experimental)
  Interventions: Drug: LAS41005
- LAS106521 (Active Comparator)
  Interventions: Drug: LAS106521
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Placebo Gel — Topical
  Arms: Placebo
Drug: LAS41005 — Topical
  Arms: LAS41005
Drug: LAS106521 — Topical
  Arms: LAS106521

SUMMARY:
The purpose of this study is to investigate the efficacy of LAS41005 in comparison to placebo and to LAS106521 in actinic keratosis (AK).

DETAILED DESCRIPTION:
To investigate as primary objective:

* Superiority to placebo and non-inferiority to LAS106521 measured by histological clearance of one predefined target lesion;

To investigate as secondary objective:

* Superiority to LAS106521
* Improvement of treated lesions (lesion response)
* Assessment of tolerability and safety by physicians global assessment score (PGA, PGT)
* Patient's assessment of tolerability and efficacy and patient's compliance

ELIGIBILITY:
Main Inclusion Criteria:

* Have at least 4 but not more than 10 clinically confirmed AK target lesions of mild to moderate intensity within the face/forehead or bald scalp (excluding eyelids, lips, and mucosa), i.e. actinic keratosis grade I and II according to Olsen EA et al. 1991
* Woman of childbearing potential are allowed to participate in this study only if they use a highly effective method of contraception

Main Exclusion Criteria:

* Have received effective treatment of AK in the three months preceding this clinical trial
* Have known hypersensitivity to LAS41005 or LAS106521
* Have currently other malignant or benign tumors of the skin within the treatment area (e.g. malignant melanoma, basal cell carcinoma, squamous cell carcinoma)
* Patient's taking phenytoin
* Show cornu cutaneum like alterations of the skin in the face or the bald scalp (target area)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Histological status of AK target lesion | Day 140

CONTACTS AND LOCATIONS:
Overall Officials: Estrella Garcia, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (40):
- Germany (40):
  - Almirall Facility Site#37, Altenkirchen
  - Almirall Facility Site#24, Augsburg
  - Almirall Facility Site#23, Augsburg
  - Almirall Facility Site#01, Berlin
  - Almirall Facility Site#28, Berlin
  - Almirall Facility Site#02, Berlin
  - Almirall Facility Site#34, Berlin
  - Almirall Facility Site#35, Berlin
  - Almirall Facility Site#31, Bonn
  - Almirall Facility Site#04, Buxtehude
  - Almirall Facility Site#40, Detmold
  - Almirall Facility Site#30, Dresden
  - Almirall Facility Site#11, Dülmen
  - Almirall Facility Site#12, Düsseldorf
  - Almirall Facility Site#17, Frankfurt
  - Almirall Facility Site#22, Freiburg im Breisgau
  - Almirall Facility Site#36, Friedrichshafen
  - Almirall Facility Site#19, Fulda
  - Almirall Facility Site#32, Göttingen
  - Almirall Facility Site#09, Hamburg
  - Almirall Facility Site#29, Jena
  - Almirall Facility Site#07, Kiel
  - Almirall Facility Site#08, Kiel
  - Almirall Facility Site#15, Koblenz
  - Almirall Facility Site#21, Landau
  - Almirall Facility Site#27, Leipzig
  - Almirall Facility Site#06, Lübeck
  - Almirall Facility Site#03, Mahlow
  - Almirall Facility Site#25, München
  - Almirall Facility Site#39, München
  - Almirall Facility Site#33, Nördlingen
  - Almirall Facility Site#38, Osnabrück
  - Almirall Facility Site#05, Pinneberg
  - Almirall Facility Site#26, Quedlinburg
  - Almirall Facility Site#20, Radolfzell
  - Almirall Facility Site#10, Salzwedel
  - Almirall Facility Site#16, Soest
  - Almirall Facility Site#14, Vechta
  - Almirall Facility Site#18, Wiesbaden
  - Almirall Facility Site#13, Wuppertal

REFERENCES:
- See also: Sponsor website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp